CLINICAL TRIAL: NCT07222943
Title: Open-Labelled Feasibility Study of a Guided Imagery Therapy Mobile Application for Functional Abdominal Pain Disorders in Children
Brief Title: Feasibility Study of a Guided Imagery Therapy Mobile Application for Functional Abdominal Pain Disorders in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, John M Hollier, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-58306
Record Dates: First submitted 2025-10-26; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Functional Abdominal Pain Disorders; Irritable Bowel Syndrome (IBS); Functional Gastrointestinal Disorders (FGIDs); Gastrointestinal and Digestive Disorder; Abdominal Pain/ Discomfort; Pain; Functional Dyspepsia
Keywords: abdominal pain; irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases; Digestive System Diseases; Pain; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: Qualified participants will be given access to the mobile app intervention for eight weeks. At the end of the eight weeks, outcome measures will be reassessed through an abdominal pain and stooling diary and other surveys. we will also assess these same outcomes 3 months -post-treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants randomized to the Immediate Treatment arm will receive immediate access to the guided imagery therapy mobile application intervention.
  Interventions: Behavioral: Guided Imagery Therapy

INTERVENTIONS:
Behavioral: Guided Imagery Therapy — Participants will be asked to listen to a pre-recorded, 10 to 15 minute guided imagery therapy (GIT) sessions via mobile application 5 out of 7 days per week for 8 weeks in addition to their usual care for their abdominal pain.

SUMMARY:
Chronic abdominal pain is common among children, and the majority of cases are attributed to functional abdominal pain disorders. One approach to treating these disorders is by using psychological therapies. This clinical trial aims to see how well pre-recorded guided imagery therapy sessions help children's abdominal pain when delivered via a mobile application (app) on a smartphone or tablet.

Participants will complete a baseline abdominal pain and stooling diary to determine eligibility, as well as other surveys. Eligible participants will be given access to the guided imagery therapy mobile application.

This intervention asks participants to listen to a 10- to 15-minute GIT session 5 out of 7 days per week for 8 weeks, in addition to their usual care for their abdominal pain. Then, participants will complete another abdominal pain and stooling diary, along with other psychometric surveys, at the end of this intervention period. Participants will also collect another diary and surveys 3 months post-treatment.

DETAILED DESCRIPTION:
After fully disclosing the study design, intervention options, randomization scheme, and potential side effects of the interventions, caregivers and their children will document their respective informed consent and assent electronically. REDCap is a secure web application designed for surveys and databases. All data captured through REDCap will be encrypted and transmitted securely to HIPAA-compliant institutional servers for storage.

Participants and their caregivers will complete the following surveys at baseline, immediately post-therapy (8 weeks after baseline), and 3 months post-treatment through REDCap:

* 2-week Abdominal Pain and Stooling Diary
* Children's Somatic Symptoms Inventory (child self-report and parent proxy-report)
* Pain Catastrophizing Scale - Child Version
* Pain Catastrophizing Scale - Parent Version
* Pediatric Quality of Life Inventory 4.0 Generic Core (child self-report and parent proxy-report)
* Behavior Assessment System for Children 3rd Ed (child self-report and parent proxy-report)

ELIGIBILITY:
Inclusion Criteria:

* Texas Children's Pediatrics patients 7 to 12 years old at enrollment
* A Rome IV Functional Abdominal Pain Disorder as defined by a 2-week abdominal pain and stooling diary
* Both children and their primary caregivers must be able to read and communicate in English proficiently to understand the intervention's audio therapy sessions and psychometric instruments.

Exclusion Criteria:

* Previous abdominal surgeries
* Co-morbid conditions associated with abdominal pain (e.g., cystic fibrosis)
* Autism
* Significant development delay
* Psychosis
* Prior experience with cognitive behavioral therapy or guided imagery therapy to treat chronic abdominal pain
* Alarm symptoms that warrant further medical evaluation (e.g., blood in stool)

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Abdominal Pain Intensity | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Average daily abdominal pain severity measured on a 0-10 (10 is most severe) ordinal scale from a self-report 2-week abdominal pain diary

SECONDARY OUTCOMES:
Abdominal Pain Frequency | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Average number of abdominal pain episodes per day from a self-report 2-week abdominal pain diary
Anxiety | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Behavior Assessment System for Children, third edition, child self-report Anxiety Scale, t score ranges from 20 to 120, higher scores are worse
Anxiety | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Behavior Assessment System for Children, third edition, parent proxy-report Anxiety Scale, t score ranges from 20 to 120, higher scores are worse
Depression | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Behavior Assessment System for Children, third edition, child self-report Depression scale, t score ranges from 20 to 120, higher scores are worse
Depression | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Behavior Assessment System for Children, third edition, parent-proxy report Depression scale, t scores ranges from 20 to 120, higher scores are worse
Somatization | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Children's Somatic Symptoms Inventory child self-report, raw score ranges from 0 to 96, higher scores are worse
Somatization | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Children's Somatic Symptoms Inventory parent-proxy report, raw score ranges from 0 to 96, higher scores are worse
Pain Catastrophizing Thoughts | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Pain Catastrophizing Scale - Child Version, raw score ranges from 0 to 52, higher scores are worse
Pain Catastrophizing Thoughts | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Pain Catastrophizing Scale - Parent Version, raw score range from 0 to 52, higher scores are worse
Health-Related Quality of Life | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Pediatric Quality of Life Inventory Generic Core Scales 4.0 child self-report, raw score ranges from 0 to 100, higher scores are better
Health-Related Quality of Life | Baseline, Post-intervention (immediately after 8-week intervention), and 3-months Post-Treatment
  Pediatric Quality of Life Inventory Generic Core Scales 4.0 parent-proxy report, raw score ranges from 0 to 100, higher scores are better

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baylor College of Medicine/Texas Children's Hospital, Austin, Texas
  - Baylor College of Medicine / Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided